CLINICAL TRIAL: NCT06223802
Title: Balance Response to Biodex Training in Hemodialysis Females With Osteopenia
Brief Title: Biodex Training in Hemodialysis Females With Osteopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Hagar Ahmed El-Hadidy, lecturer of physical therapy for Internal Medicine and Geriatrics, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004928
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Hemolysis
MeSH Terms: conditions — Hemolysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trained group (Experimental): women group with a number of 29 women receiving 3-time biodex training per week, every time will be 10 minutes for 12 weeks
  Interventions: Behavioral: biodex training
- non trained group (No Intervention): this group will serve as a control group that will receive no intervention

INTERVENTIONS:
Behavioral: biodex training — women group with a number of 29 women receiving 3-time biodex training per week, every time will be 10 minutes for 12 weeks
  Arms: trained group

SUMMARY:
imbalance is a common problem in hemodialysis patients with osteopneia, biodex training is a good device that treat imbalance

DETAILED DESCRIPTION:
58 women with osteopenia problem and dialysis will be divided to trained women group with a number of 29 women receiving 3-time biodex training per week, every time will be 10 minutes for 12 weeks or nontrained women group that will act as a control group (n = 29 women)

ELIGIBILITY:
Inclusion Criteria:

* osteopneia women
* hemodialysis women

Exclusion Criteria:

* pregnancy
* autoimmune disorders
* lower limb orthopedic problems
* psychological manifestaion

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 58 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-03-08 (Estimated); Study Completion 2024-03-08 (Estimated)

PRIMARY OUTCOMES:
bone mineral density of femur bone | it will be measured after 12 weeks
  it will be measured by DEXA

SECONDARY OUTCOMES:
overall stability index | it will be measured after 12 weeks
  it a parameter indicates the good balance of patients
Antero posterior stability index | it will be measured after 12 weeks
  it a parameter indicates the good balance of patients
Mediolateral stability index | it will be measured after 12 weeks
  it a parameter indicates the good balance of patients
six minute walk test | it will be measured after 12 weeks
  it a parameter asses funntional capacity
Short physical performance battery | it will be measured after 12 weeks
  total score or points will be assessed from this physical performance test

CONTACTS AND LOCATIONS:
Overall Officials: hagar El-Hadidy, lecturer, Principal Investigator — Ahram Canadian University
Locations (1):
- Ahram canadian university, Giza, Egypt